CLINICAL TRIAL: NCT07275411
Title: Tele-education Through a New Mobile Application to Improve Oral Cancer Knowledge and Oral Hygiene in Older Adults
Brief Title: mHealth App for Oral Hygiene and Cancer Awareness in Older Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Chile (Other)
Collaborators: Universidad de La Frontera (Other)
Responsible Party: Principal Investigator, Iris Espinoza Santander, Associate Professor, University of Chile
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: CIES009
Record Dates: First submitted 2025-11-27; First posted 2025-12-10 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-06

CONDITIONS: Oral Cancer; Oral Health Knowledge, Attitude and Practice Among Patients; Older Adults
MeSH Terms: conditions — Mouth Neoplasms; Behavior

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Serious Games Group (Experimental): Participants receive an oral health mobile application with educational videos and serious games designed to improve knowledge and self-examination practices.
  Interventions: Behavioral: Mobile Oral Health Education App
- Video-Only Group (Active Comparator): Participants receive an oral health mobile application with educational videos only, without interactive components.
  Interventions: Behavioral: Mobile Oral Health Education App

INTERVENTIONS:
Behavioral: Mobile Oral Health Education App — This intervention consists of a mobile application designed to improve oral health knowledge, attitudes, and practices among older adults. The app includes educational videos about oral hygiene and oral cancer. In the experimental group, the app also incorporates interactive serious games to reinforce learning and promote oral self-examination. In the active comparator group, participants have access only to the educational videos within the same app. The intervention targets individuals aged 60 to 70 years and is evaluated over a 4-week period through questionnaires and observation of oral self-examination practices.

SUMMARY:
The goal of this clinical trial is to learn whether a mobile app with educational videos and serious games is more effective than a video-only version of the app to improve knowledge, attitudes, and practices about oral cancer and oral hygiene in older adults.

The study also aims to evaluate the usability of the app and the impact of the intervention on performing oral self-examination.

The main questions it aims to answer are:

1. - Does the version of the app with videos and serious games lead to greater improvement in oral cancer knowledge than the video-only version?
2. - Are there differences in attitudes and self-examination practices between the two groups after using the app?
3. - How frequently and consistently do participants use the app during the study period, and how much do they interact with the educational videos and serious games?
4. - Are there differences in outcomes by sex or education level?

Participants will:

Be adults aged 60 and more receiving care at the Dental Clinic of the University of Chile

Be randomly assigned to use one of two versions of the same app:

* Group A: Access to educational videos and serious games
* Group B: Access to educational videos only

Use the app for 4 weeks

Answer a questionnaire before starting, after 2 weeks, and after 4 weeks

Perform an oral self-examination at week 4, which will be evaluated using a checklist

This trial will help determine whether mobile tele-education tools, especially those that include interactive features like serious games, are effective and acceptable ways to improve oral health education in older adults.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 60 years and older.
* Completed dental treatment at the Dental Clinic of the Faculty of Dentistry, University of Chile, during 2023 and 2024.
* Own a smartphone with Android operating system.
* Regular users of at least one social media platform (e.g., WhatsApp, Instagram, Facebook).

Exclusion Criteria:

* Older adults with self-reported uncorrected visual or auditory sensory deficits resulting in total blindness or deafness.
* Older adults with cognitive impairment, defined as a score of 13 or lower on the abbreviated Mini-Mental State Examination (MMSE) (maximum score 19).

Ages: 60 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2024-05-02 (Actual); Primary Completion 2024-11-11 (Actual); Study Completion 2024-11-11 (Actual)

PRIMARY OUTCOMES:
Change in knowledge, attitudes about oral cancer and oral hygiene, and performance of oral self-examination in older adults using a mobile educational application. | Baseline, 2 weeks, and 4 weeks after the start of the intervention.
  increasing participants' knowledge and attitudes regarding oral cancer and oral hygiene, as well as their ability to perform oral self-examination. Knowledge and attitudes are measured using a structured questionnaire administered at baseline, 2 weeks, and 4 weeks. Oral self-examination practices are evaluated at 4 weeks using a standardized checklist verifying the correct performance of five key steps. Comparisons are made between the group using videos and serious games and the group using videos only.

SECONDARY OUTCOMES:
Usability of the mobile oral health education application | 4 weeks
  Evaluates participant use and engagement with the mobile app by analyzing interaction logs recorded within the app over the 4-week intervention period. Usage data are compared between the group using videos plus serious games and the group using videos only.

CONTACTS AND LOCATIONS:
Overall Officials: Iris Lucia Espinoza-Santander, PhD in Public Health, Principal Investigator — Departament of Pathology and Oral Medicine, Faculty of Dentistry, University of Chile; Constanza Beatriz Morales-Gómez, Master's Degree in Science, Study Chair — Departament of Pathology and Oral Medicine, Faculty of Dentistry, University of Chile
Locations (1):
- Dental Clinic, Faculty of Dentistry, University of Chile, Santiago, Chile